CLINICAL TRIAL: NCT00173550
Title: Perception and Attitude Toward Estrogen Therapy Among Operated Women With Premature or Immature Menopause
Brief Title: Perception and Attitude Toward Estrogen Therapy Among Surgically Menopausal Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: 9461700710; NSC93-2314-B-002-162
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-01-23 (Estimated); Status verified 2005-07

CONDITIONS: Menopause, Premature; Hysterectomy; Ovariectomy; Estrogen Replacement Therapy; Attitude; Perception
Keywords: Menopause, premature; Hysterectomy; Ovariectomy; Estrogen Replacement Therapy; Knowledge; Perception; Attitude
MeSH Terms: conditions — Menopause, Premature; Behavior | interventions — Hysterectomy

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Procedure: Hysterectomy and Bilateral salpingo-oophorectomy

SUMMARY:
The aim of this study is to survey patient's cognition and attitude about health-related quality of life, use of estrogen, experience of menopausal syndrome, compliance of medication, experience, and satisfaction for women who underwent hysterectomy and bilateral oophorectomy before menopause.

DETAILED DESCRIPTION:
The cognition and attitude of menopausal women toward hormone replacement could have been changed since the report from WHI in July 2002. Previously, many women used hormone replacement to prevent cardiovascular disease and osteoporosis. Recently, the use has been challenged, exaggerated, and also discussed both in media press and academic meetings. Many women dare not to use them. The women who underwent hysterectomy and bilateral salpingo-oophorectomy before menopause may immediately face the problems caused by deficiency of female sex hormone. For this group of women, as yet there is no conclusion about whether the women should take hormone replacement therapy for a long time to osteoporosis, cardiovascular disease and other chronic disease. The arm for this study from WHI is not closed yet. While the women in our area might have been influenced by this report and have changed their mind. It is essential for us to make a clear understanding about the cognition and attitude for hormone replacement therapy for women who underwent hysterectomy and bilateral salpingo- oophorectomy. Therefore, it may be a pioneer study and worthwhile to do this study. Data from a medical center from 2000 to 2004 will be examined for evidence of bilateral oophorectomy & hysterectomy. The cause for the surgery will be confirmed by pathological findings. These women who were under 50 years of age will be candidate of the study. The women will be interviewed about their beliefs, and cognition, regarding their quality of life and health risks as well as their opinion on menopause and hormone replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age under 50
* Hysterectomy and bilateral oophorectomy

Exclusion Criteria:

* Unwilling to answer the questionnaires

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200
Dates: Start 2004-08

CONTACTS AND LOCATIONS:
Overall Officials: Ruey-Jien Chen, MD, PhD, Principal Investigator — Department or Obstetrics and Gynecology, National Taiwan university Hospital
Locations (1):
- National Taiwan University Hospital Department of Obstetrics and Gynecology, Taipei, Taipei, Taiwan

REFERENCES:
- [Background] Anderson GL, Limacher M, Assaf AR, Bassford T, Beresford SA, Black H, Bonds D, Brunner R, Brzyski R, Caan B, Chlebowski R, Curb D, Gass M, Hays J, Heiss G, Hendrix S, Howard BV, Hsia J, Hubbell A, Jackson R, Johnson KC, Judd H, Kotchen JM, Kuller L, LaCroix AZ, Lane D, Langer RD, Lasser N, Lewis CE, Manson J, Margolis K, Ockene J, O'Sullivan MJ, Phillips L, Prentice RL, Ritenbaugh C, Robbins J, Rossouw JE, Sarto G, Stefanick ML, Van Horn L, Wactawski-Wende J, Wallace R, Wassertheil-Smoller S; Women's Health Initiative Steering Committee. Effects of conjugated equine estrogen in postmenopausal women with hysterectomy: the Women's Health Initiative randomized controlled trial. JAMA. 2004 Apr 14;291(14):1701-12. doi: 10.1001/jama.291.14.1701. PMID 15082697
- [Background] Levens E, Williams RS. Current opinions and understandings of menopausal women about hormone replacement therapy (HRT)-the University of Florida experience. Am J Obstet Gynecol. 2004 Aug;191(2):641-6; discussion 646-7. doi: 10.1016/j.ajog.2004.06.074. PMID 15343254
- See also: library of National taiwan University Hospital — http://ntuml.mc.ntu.edu.tw